CLINICAL TRIAL: NCT00388440
Title: Phase IV Open Study to Assess the Safety, Reactogenicity and Immunogenicity of GlaxoSmithKline (GSK) Biologicals' Live Attenuated Measles-Mumps-Rubella (MMR) Vaccine When Given to Healthy Children at the Age of 12 to 18 Months in Singapore.
Brief Title: Assess GSK Biologicals' MMR Vaccine (Priorix) When Given to Healthy Children at the Age of 12 to 18 Months in Singapore.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 209762/147
Record Dates: First submitted 2006-10-13; First posted 2006-10-16 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Rubella; Mumps; Measles
Keywords: Mumps; Singapore; Rubella; Measles
MeSH Terms: conditions — Rubella; Mumps; Measles | interventions — Measles-Mumps-Rubella Vaccine

INTERVENTIONS:
Biological: MMR vaccine (Priorix)

SUMMARY:
To evaluate the safety and immunogenicity of GSK Biologicals' live attenuated MMR vaccine (Priorix) in a local population in Singapore. The vaccine was administered as a single dose to healthy children (12-18 months of age) and blood samples were collected at two time points (before vaccination and after vaccination).

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant between 12 and 18 months of age at the time of the vaccination
* Written informed consent obtained from the parents or guardians of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) during the study period or within 30 days preceding the dose of study vaccine
* Previous vaccination against mumps and/or rubella
* History of, or intercurrent, measles, mumps, and/or rubella disease
* Known exposure to measles, mumps or rubella within 30 days prior to the start of the study
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2000-11; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Solicited symptoms (Day 0-3); unsolicited AEs (Day 0-42); SAEs (full study)

SECONDARY OUTCOMES:
Antibody concentration to all vaccine antigens after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 209762/147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 209762/147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 209762/147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 209762/147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 209762/147 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register